CLINICAL TRIAL: NCT00717132
Title: Cost-effectiveness of Family Based Pediatric Obesity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Healthnow (Unknown)
Responsible Party: Principal Investigator, Leonard Epstein, Leonard H. Epstein, Ph.D., State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cost-effectiveness; A-45270 (Other Grant/Funding Number: HealthNow)
Record Dates: First submitted 2008-07-10; First posted 2008-07-16 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Weight Change; Quality of Life
Keywords: weight; cost effectiveness; obesity; family based behavioral treatment
MeSH Terms: conditions — Body Weight Changes; Body Weight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual Behavioral Modification (Experimental): Individual behavioral weight control treatment; parent and child are treated separately for 15 total sessions.
  Interventions: Behavioral: Individual Behavior Modification
- Family-based Behavioral Modification (Active Comparator): Family-based behavioral weight control treatment; parent and child are treated together for 15 total sessions.
  Interventions: Behavioral: Family-based behavior modification

INTERVENTIONS:
Behavioral: Individual Behavior Modification — Individual behavioral treatment for obesity. Children and parents meeting individually for 15 total behavioral modification intervention sessions.
  Arms: Individual Behavioral Modification
Behavioral: Family-based behavior modification — Family-base behavior treatment for obesity. Children and parents meeting together for 15 total behavioral modification intervention sessions.
  Arms: Family-based Behavioral Modification

SUMMARY:
To determine the cost effectiveness of treating the child alone and parent alone to traditional family-based method of obesity treatment. It is hypothesized that a family-based approach will be more cost effective, and will support the savings and effectiveness of treating multiple family members together.

DETAILED DESCRIPTION:
Research has shown that family-based treatment programs produce significant short and long-term decreases in weight relative to height. Reductions in relative weight are observed for both parents and their children, with a significant relationship between parent and child relative weight changes.

Usual care for families with obesity is for the parent and child to be treated separately by their individual physicians, often with different types of treatment plans. This may be less efficacious for the parent and child than a family-based intervention in which the parent and child are treated together. The separate treatments may also be more expensive than concurrent treatment following the same treatment plan.

There are many reasons to hypothesize that a family-based treatment will be more efficacious and more cost effective than other formats for treating families with multiple generations of obesity. If family members are treated together, they have the same treatment goals. They can learn to support each other, model positive behaviors, work together to change behaviors and modify the shared family environment. The simultaneous treatment of parents and children in a group format, which is how family-based treatments are administered, reduces the time therapists provide treatment in comparison to the usual format in which each parent and child would be seen individually.

An important challenge for obesity treatment is to develop efficacious and cost-effective interventions to treat pediatric obesity. The goal of this study is to evaluate the efficacy and cost effectiveness over 12 month follow-up for 50 families with overweight parents and children randomized to family-based behavioral treatment in comparison to the treatment of the parents and children separately, by different therapists, which represent usual care for families with obese parents and children.

ELIGIBILITY:
Inclusion Criteria:

* Overweight child and parent in each family

Exclusion Criteria:

* The parent and child must have no dietary or activity limitations that would preclude making the requested behavior changes; no current psychiatric problems and no history of eating disorders, including anorexia nervosa, bulimia nervosa or binge eating disorder. Families with a first degree relative with any of the mentioned eating disorders will also be excluded. The participating child must be able to read at a 3rd grade level and demonstrate the ability to maintain diet and activity records in a simulated recording interview. Both parent and child must be able to read the English language well enough to understand the consent and assent forms.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in Standardized BMI | baseline, 6 months, 12 months
  The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared. Children's BMI also accounts for age and sex.

SECONDARY OUTCOMES:
change in quality adjusted life years (QALY) | baseline, 6 months, 12 months
  The quality-adjusted life-year (QALY) is a measure of the value of health outcomes. Health is calculated by length of life and quality of life. QALY takes the value of years living and the quality into a single index number. The QALY calculation is the change in utility value resulting from the treatment multiplied by the duration of the treatment effect to provide the number of QALYs. QALYs can then be incorporated with medical costs to arrive at a final common denominator of cost/QALY.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H Epstein, PhD, Principal Investigator — SUNY @ Buffalo
Locations (1):
- SUNY @ Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted